CLINICAL TRIAL: NCT00551213
Title: A Fixed-Sequence, Open-Label Study to Determine the Activity of SCH 717454 as Assessed by Positron Emission Tomography in Subjects With Relapsed or Recurrent Colorectal Cancer
Brief Title: A Study to Determine the Activity of Robatumumab (SCH 717454, MK-7454) in Participants With Relapsed or Recurrent Colorectal Cancer (P04721, MK-7454-003)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P04721; MK-7454-003 (Other: Merck Protocol Number)
Record Dates: First submitted 2007-10-29; First posted 2007-10-30 (Estimated); Results first posted 2015-12-15 (Estimated); Last update posted 2018-08-24 (Actual); Status verified 2018-07

CONDITIONS: Colorectal Cancer
Keywords: anti-IGF-1R
MeSH Terms: conditions — Colorectal Neoplasms | interventions — robatumumab; Irinotecan; Cetuximab; Capecitabine; Folfox protocol; XELOX; IFL protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Robatumumab→Robatumumab (Experimental): Participants receive 1 dose of robatumumab 0.3 mg/kg intravenously (IV) followed by 1 dose of robatumumab 10 mg/kg IV once every 2 weeks (Q2W) until disease progression. A cycle of robatumumab is defined as 2 weeks of treatment (i.e., 1 dose of robatumumab) with no recovery period between cycles.
  Interventions: Biological: Robatumumab
- Chemotherapy→Robatumumab (Active Comparator): Participants receive 1 cycle of standard colorectal cancer chemotherapy currently approved and available on the market for use in colorectal cancer (to be selected by the Investigator based on participant's prior treatment) followed by 1 dose of robatumumab 10 mg/kg IV Q2W until disease progression. A cycle of robatumumab is defined as 2 weeks of treatment (i.e., 1 dose of robatumumab) with no recovery period between cycles.
  Interventions: Biological: Robatumumab; Drug: Irinotecan; Biological: Cetuximab; Drug: Capecitabine; Drug: FOLFOX; Drug: CAPEOX/XELOX; Drug: FOLFIRI

INTERVENTIONS:
Biological: Robatumumab
Drug: Irinotecan
  Arms: Chemotherapy→Robatumumab
Biological: Cetuximab
  Arms: Chemotherapy→Robatumumab
Drug: Capecitabine
  Arms: Chemotherapy→Robatumumab
Drug: FOLFOX — Leucovorin calcium (folinic acid)(FOL) + 5-fluorouracil (F)+ oxaliplatin (OX)
  Arms: Chemotherapy→Robatumumab
Drug: CAPEOX/XELOX — Capecitabine (CAPE) or Xeloda® (XEL) + oxaliplatin (OX)
  Arms: Chemotherapy→Robatumumab
Drug: FOLFIRI — Leucovorin calcium (folinic acid)(FOL) + 5-fluorouracil (F)+ irinotecan (IRI)
  Arms: Chemotherapy→Robatumumab

SUMMARY:
The purpose of this study was to determine the activity of two doses of robatumumab (SCH 717454, MK-7454) in participants with relapsed or recurrent colorectal cancer.

The primary study hypothesis was that decreases in Positron Emission Tomography (PET)-assessed tumor glucose metabolism (i.e., fluorodeoxyglucose [FDG] standardized uptake value [SUV]) following administration of 10 mg/kg robatumumab will exceed those following administration of 0.3 mg/kg robatumumab in participants with relapsed or recurrent colorectal cancer who had progressed after first-line chemotherapy.

Investigator choices of standard chemotherapy: irinotecan as a single agent +/- cetuximab OR capecitabine as a single agent, OR FOLFOX (leucovorin calcium [folinic acid][FOL] + fluorouracil [F] + oxaliplatin [OX]) OR CAPEO(capecitabine [CAPE] or Xeloda® [XEL] + oxaliplatin [OX]) OR FOLFIRI (leucovorin calcium [folinic acid][FOL] + fluorouracil [F] + irinotecan [IRI]) +/- cetuximab OR cetuximab as a single agent.

DETAILED DESCRIPTION:
Standard chemotherapy was used as a positive validation arm. Randomization was performed so that there could be no bias in the selection of participants for enrollment into the fixed-sequence arms. Once three chemotherapy-treated participants demonstrated decreases in FDG-PET SUV in the target lesion (i.e., >20% decrease in SUVmax in the defined target lesion) in the PET/computed tomography (CT) scan performed following Cycle 1 Period 1 treatment, it was concluded that this positive validation arm had accomplished its purpose, and all subsequent participants enrolled in the study were assigned treatment with robatumumab for Period 1. There was no intention to compare the data in either period across participants who received chemotherapy with those who received robatumumab.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years of age, of any race, and gender;
* Diagnosis of histologically confirmed relapsed or recurrent colorectal carcinoma that has progressed on at least first-line therapy;
* Must have a computed tomography (CT) or magnetic resonance imaging (MRI) scan performed at some point during their immediate prior treatment or observation in order to determine tumor growth rate;
* Must have measurable disease on a CT or MRI study, performed during Screening;
* Must have an Eastern Cooperative Oncology Group (ECOG) performance status of <=2 and a minimum life expectancy of ≥4 months;
* Must have adequate organ function within 3 weeks prior to treatment assignment

Exclusion Criteria:

* History of another malignancy;
* Known treated or untreated leptomeningeal metastasis, or a metastatic central nervous system lesion;
* Surgery within 3 weeks;
* Radiation therapy within 6 weeks;
* A history of uncontrolled diabetes mellitus, defined as a hemoglobin A1C of >7.5% in a participant with known diabetes mellitus;
* A recent myocardial infarction (within the past year); or a participant who at the time of Screening presents with unstable or uncontrolled angina, New York Heart Association Class III or IV congestive heart failure, uncontrolled hypertension, clinically significant cardiac dysrhythmia or clinically significant electrocardiogram abnormality;
* An active infection;
* Has clinically significant hepatitis at Screening, or is hepatitis C antibody positive, hepatitis B surface antigen positive, or human immunodeficiency virus (HIV) seropositive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2007-11-21 (Actual); Primary Completion 2009-06-04 (Actual); Study Completion 2009-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Lin EH, Lenz HJ, Saleh MN, Mackenzie MJ, Knost JA, Pathiraja K, Langdon RB, Yao SL, Lu BD. A randomized, phase II study of the anti-insulin-like growth factor receptor type 1 (IGF-1R) monoclonal antibody robatumumab (SCH 717454) in patients with advanced colorectal cancer. Cancer Med. 2014 Aug;3(4):988-97. doi: 10.1002/cam4.263. Epub 2014 Jun 6. PMID 24905030
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=P04721&kw=P04721&tab=access

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Robatumumab→Robatumumab | Chemotherapy→Robatumumab
Started | 50 | 17
Treated | 49 | 15
Completed | 0 | 0
Not Completed | 50 | 17
Not completed — Adverse Event | 6 | 3
Not completed — Progressive Disease | 41 | 12
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Not Treated | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Robatumumab→Robatumumab: Participants receive 1 dose of robatumumab 0.3 mg/kg IV followed by 1 dose of robatumumab 10 mg/kg IV Q2W until disease progression. A cycle of robatumumab is defined as 2 weeks of treatment (i.e., 1 dose of robatumumab) with no recovery period between cycles.
- Total: Total of all reporting groups
Arm/Group | Robatumumab→Robatumumab | Chemotherapy→Robatumumab | Total
Number analyzed (Participants) | 50 | 17 | 67
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.7 (10.8) | 61.9 (10.6) | 64.0 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 9 | 39
  Male | 20 | 8 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a >20% Decrease in Positron Emission Tomography (PET)-Assessed Tumor Glucose Metabolism: Fluorodeoxyglucose (FDG) Standardized Uptake Value (SUV) in the Target Lesion
Description: FDG-PET was used in this study to detect the biological activity of modulation of the target within the tumor. Response Evaluation Criteria in Solid Tumors (RECIST) version 1.0 was used to select the target lesion. All measurable lesions up to a maximum of 5 lesions per organ and 10 lesions in total, representative of all involved organs were identified as target lesions and recorded and measured at Baseline. The changes in SUVmax were calculated using the formula: (endpoint SUVmax - baseline SUVmax)/baseline SUVmax as a percentage. If multiple lesions had been measured at a visit, percentages calculated for all target lesions were averaged to find the decrease during the treatment period per participant. FDG SUVmax responder was defined as participants with >20% decrease in SUVmax after the first cycle of robatumumab in Period 2.
Time Frame: After the first robatumumab dose in Period 2 (Up to approximately 4 weeks after first robatumumab dose in Period 1)
Population: All participants who received ≥1 dose of robatumumab in Periods 1 and 2 and had SUV data before and after the first dose of robatumumab in Period 2 were included in the analysis. No participants in the Chemotherapy→Robatumumab group received robatumumab in Period 1.
Measure: Number; unit: Participants
Arm/Group | Robatumumab→Robatumumab | Chemotherapy→Robatumumab
Number analyzed (Participants) | 41 | 0
Participants | 7 [7 to 32] |

2. Secondary Outcome: Number of Participants Who Experienced One or More Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant administered study drug which does not necessarily have a causal relationship with the study drug. AEs may include the onset of new illness and the exacerbation of pre-existing conditions.
Time Frame: Up to 30 days after last dose of study drug (Up to approximately 22 weeks)
Population: All participants who received ≥1 dose of study drug were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Robatumumab→Robatumumab | Chemotherapy→Robatumumab
Number analyzed (Participants) | 49 | 15
Participants | 49 | 15

3. Secondary Outcome: Best Overall Tumor Response Per Investigator Review
Description: Tumor response was assessed by computed tomography (CT) or magnetic resonance imaging (MRI) scans using RECIST v 1.0 criteria at Screening, at every 8 weeks of robatumumab treatment during Period 2 and at post study. A sum of the longest diameter (LD) for all target lesions was calculated and reported as the baseline sum LD. Overall tumor responses were defined as: Complete Response (CR) - Disappearance of all target lesions; Partial Response (PR) - At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD; Progressive Disease (PD) - At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; or Stable Disease (SD) - Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: Up to 30 days after last dose of study drug (Up to approximately 22 weeks)
Population: All participants who received ≥1 dose of robatumumab were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Robatumumab→Robatumumab | Chemotherapy→Robatumumab
Number analyzed (Participants) | 49 | 15
Participants
  Partial Response | 1 | 0
  Stable Disease | 10 | 7
  Progressive Disease | 33 | 6
  No post-Baseline assessment | 5 | 2

4. Secondary Outcome: Number of Participants Who Discontinued Study Drug Due to an AE
Description: as for outcome 2
Time Frame: Up to last dose of study drug (Up to approximately 18 weeks)
Population: All participants who received ≥1 dose of study drug were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Robatumumab→Robatumumab | Chemotherapy→Robatumumab
Number analyzed (Participants) | 49 | 15
Participants | 6 | 3

5. Secondary Outcome: Best Overall Tumor Response Per Central Review
Description: Tumor response was assessed by CT or MRI scan using RECIST v1.0 criteria at Screening, at every 8 weeks of robatumumab treatment during Period 2 and at post study. A sum of the LD for all target lesions was calculated and reported as the baseline sum LD. Overall tumor responses were defined as: Complete Response (CR) - Disappearance of all target lesions; Partial Response (PR) - At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD; Progressive Disease (PD) - At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; or Stable Disease (SD) - Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: Up to 30 days after last dose of study drug (Up to approximately 22 weeks)
Population: All participants who received ≥1 dose of robatumumab were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Robatumumab→Robatumumab | Chemotherapy→Robatumumab
Number analyzed (Participants) | 49 | 15
Participants
  Partial Response | 0 | 0
  Stable Disease | 10 | 5
  Progressive Disease | 31 | 9
  No post-Baseline assessment | 8 | 1

6. Secondary Outcome: Change From Baseline in Tumor Growth Rate
Description: Tumor growth rate was assessed by CT or MRI scans using RECIST criteria at Screening, at every 8 weeks of robatumumab treatment and at post study. For Pre Baseline 1, tumor growth rate=(sum of longest diameter of target lesions at Baseline - the most recent prior to Baseline)/duration between Baseline and Pre Baseline. For all other cycles, tumor growth rate=(sum of longest diameter of target lesions at a cycle - Baseline)/ duration between Baseline and the cycle. The cycles presented below are relative to the first dose of robatumumab in Period 1.
Time Frame: Baseline and up to approximately 22 weeks
Population: All participants who received ≥1 dose of robatumumab in Periods 1 and 2 were included in the analysis. No participants in the Chemotherapy→Robatumumab group received robatumumab in Period 1.
Measure: Mean (Standard Deviation); unit: mm/day
Arm/Group | Robatumumab→Robatumumab | Chemotherapy→Robatumumab
Number analyzed (Participants) | 49 | 0
mm/day
  Pre Baseline 1 (n=46) | 0.49 (0.48) |
  Cycle 1 (n=24) | 0.07 (0.67) |
  Cycle 2 (n=25) | 0.41 (0.57) |
  Cycle 5 (n=25) | 0.53 (0.63) |
  Cycle 9 (n=7) | 0.19 (0.26) |

ADVERSE EVENTS:
Time Frame: Up to approximately 22 weeks
Description: All participants who received ≥1 dose of study drug. Adverse events are reported based on the study drug a participant was taking at the time of the event.
Arm/Group | Chemotherapy→Robatumumab | Robatumumab→Robatumumab
Serious Adverse Events (participants affected / at risk) | 6/15 | 14/49
Other Adverse Events (participants affected / at risk) | 15/15 | 48/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy→Robatumumab (N=15) | Robatumumab→Robatumumab (N=49)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 3 (4)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 1 (2)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 3 (4)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (2) | 0 (0)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 3 (4)
ASTHENIA (General disorders) | 0 (0) | 1 (1)
CATHETER RELATED COMPLICATION (General disorders) | 0 (0) | 1 (1)
CHEST PAIN (General disorders) | 0 (0) | 1 (1)
MALAISE (General disorders) | 0 (0) | 1 (2)
PAIN (General disorders) | 0 (0) | 1 (2)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 1 (1)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 0 (0) | 1 (1)
BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 1 (1)
KLEBSIELLA BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1)
PERIHEPATIC ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
TOOTH INFECTION (Infections and infestations) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 1 (1)
MENTAL STATUS CHANGES (Psychiatric disorders) | 1 (1) | 0 (0)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1)
CHILLS (General disorders) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 1 (2) | 0 (0)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 1 (2) | 0 (0)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy→Robatumumab (N=15) | Robatumumab→Robatumumab (N=49)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 2 (11)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (4) | 0 (0)
LYMPHOPENIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (10) | 1 (1)
EAR HAEMORRHAGE (Ear and labyrinth disorders) | 1 (1) | 0 (0)
LACRIMATION INCREASED (Eye disorders) | 1 (1) | 1 (1)
MYODESOPSIA (Eye disorders) | 1 (1) | 0 (0)
PHOTOPSIA (Eye disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 5 (6) | 15 (23)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 4 (5)
ASCITES (Gastrointestinal disorders) | 1 (1) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 6 (7) | 16 (22)
DIARRHOEA (Gastrointestinal disorders) | 8 (12) | 14 (19)
DRY MOUTH (Gastrointestinal disorders) | 1 (1) | 5 (5)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1) | 1 (1)
ERUCTATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
FLATULENCE (Gastrointestinal disorders) | 1 (1) | 0 (0)
FREQUENT BOWEL MOVEMENTS (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 1 (1) | 1 (1)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1) | 1 (1)
HAEMATOCHEZIA (Gastrointestinal disorders) | 1 (1) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 9 (12) | 24 (31)
ODYNOPHAGIA (Gastrointestinal disorders) | 1 (1) | 1 (1)
PROCTALGIA (Gastrointestinal disorders) | 0 (0) | 3 (5)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 2 (2)
RECTAL TENESMUS (Gastrointestinal disorders) | 1 (1) | 0 (0)
SALIVARY HYPERSECRETION (Gastrointestinal disorders) | 1 (1) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 3 (3) | 2 (2)
TOOTHACHE (Gastrointestinal disorders) | 1 (1) | 2 (2)
VOMITING (Gastrointestinal disorders) | 7 (9) | 16 (20)
ASTHENIA (General disorders) | 5 (6) | 8 (10)
CATHETER RELATED COMPLICATION (General disorders) | 1 (1) | 0 (0)
CATHETER SITE RASH (General disorders) | 1 (1) | 1 (1)
CHILLS (General disorders) | 1 (1) | 1 (1)
EARLY SATIETY (General disorders) | 1 (1) | 2 (2)
FATIGUE (General disorders) | 9 (11) | 26 (36)
GAIT DISTURBANCE (General disorders) | 2 (2) | 1 (1)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 (0) | 3 (3)
MUCOSAL INFLAMMATION (General disorders) | 1 (1) | 4 (4)
OEDEMA (General disorders) | 1 (1) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 3 (4) | 6 (8)
PAIN (General disorders) | 0 (0) | 3 (3)
PERFORMANCE STATUS DECREASED (General disorders) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 2 (2) | 0 (0)
ORAL HERPES (Infections and infestations) | 2 (2) | 0 (0)
TOOTH ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 2 (3) | 2 (2)
CONTUSION (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
THERMAL BURN (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
WRIST FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
BLOOD CALCIUM DECREASED (Investigations) | 1 (1) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 3 (4)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 (0) | 4 (4)
HAEMOGLOBIN DECREASED (Investigations) | 1 (1) | 1 (1)
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 1 (1) | 1 (1)
WEIGHT DECREASED (Investigations) | 4 (9) | 6 (10)
ANOREXIA (Metabolism and nutrition disorders) | 8 (10) | 15 (18)
DECREASED APPETITE (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
DEHYDRATION (Metabolism and nutrition disorders) | 4 (4) | 11 (14)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 2 (7) | 7 (9)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (6)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (4)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (7)
COGNITIVE DISORDER (Nervous system disorders) | 0 (0) | 3 (3)
DIZZINESS (Nervous system disorders) | 1 (1) | 4 (4)
DYSGEUSIA (Nervous system disorders) | 2 (2) | 3 (3)
HEADACHE (Nervous system disorders) | 2 (2) | 9 (11)
MEMORY IMPAIRMENT (Nervous system disorders) | 1 (1) | 2 (2)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 2 (2) | 4 (5)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 2 (2) | 3 (3)
SCIATICA (Nervous system disorders) | 1 (1) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 6 (6)
CONFUSIONAL STATE (Psychiatric disorders) | 1 (1) | 4 (5)
DEPRESSION (Psychiatric disorders) | 0 (0) | 5 (5)
DISORIENTATION (Psychiatric disorders) | 1 (1) | 0 (0)
INSOMNIA (Psychiatric disorders) | 2 (2) | 6 (8)
HAEMATURIA (Renal and urinary disorders) | 1 (1) | 0 (0)
MICTURITION URGENCY (Renal and urinary disorders) | 1 (1) | 0 (0)
NOCTURIA (Renal and urinary disorders) | 0 (0) | 3 (3)
POLLAKIURIA (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL VEIN THROMBOSIS (Renal and urinary disorders) | 1 (1) | 0 (0)
URETHRAL OBSTRUCTION (Renal and urinary disorders) | 1 (1) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 8 (8)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 6 (6)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
PARANASAL SINUS HYPERSECRETION (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
ALOPECIA (Skin and subcutaneous tissue disorders) | 4 (5) | 3 (3)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
NAIL DISCOLOURATION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3)
SKIN DISCOLOURATION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SKIN DISORDER (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
SKIN LESION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
FLUSHING (Vascular disorders) | 1 (2) | 0 (0)
HYPERTENSION (Vascular disorders) | 1 (1) | 3 (3)
HYPOTENSION (Vascular disorders) | 2 (2) | 1 (1)
SINUS TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 1 (1) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 (1) | 0 (0)
PITTING OEDEMA (General disorders) | 1 (1) | 1 (1)
BILE DUCT STENOSIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
JAUNDICE (Hepatobiliary disorders) | 1 (1) | 1 (3)
TINEA INFECTION (Infections and infestations) | 1 (1) | 0 (0)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
MENTAL STATUS CHANGES (Psychiatric disorders) | 1 (1) | 0 (0)
FACIAL WASTING (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the study.